CLINICAL TRIAL: NCT07078864
Title: The Effect of the Model-Based Care Decision Support System in Pediatric Intensive Care on Nurses' Decision Making and Opinions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Bedriye AK, Assoc. Prof. Dr., Abant Izzet Baysal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AİBÜ-HEM- BA-02
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Intensive Care Nurses
Keywords: Decision support system; Watson human care model; Family-centered care model; Pediatric Intensive Care

STUDY DESIGN:
Intervention Model Description: The study is a quasi-experimental and qualitative study in a single-group pre-post test model
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric Intensive Care Nurses (Other)
  Interventions: Other: Nursing Care Decision Support System

INTERVENTIONS:
Other: Nursing Care Decision Support System — Phase Two involves implementing the Nursing Care Decision Support System. Data will be collected using a Descriptive Information Form, the Nurse Decision-Making Scale (pre-test), and a Semi-Structured Interview Form to explore nurses' views. Nurses will receive two training sessions (totaling 4 hours) covering system use, importance, challenges, and solutions. Training will be held in two groups based on shift schedules. A one-week trial will follow, with the researcher answering questions and providing support via a WhatsApp group. Nurses must use the system for at least 15 days (maximum 30 days due to dissertation timeline). Fifteen days after use ends, the Nurse Decision-Making Scale (post-test) and interviews will assess the system's effectiveness and areas for improvement.

SUMMARY:
The Effect of the Model-Based Care Decision Support System in Pediatric Intensive Care on Nurses' Decision Making and Opinions

DETAILED DESCRIPTION:
This study is designed as a mixed-method research aiming to determine the effect of using a Model-Based Care Decision Support System in Pediatric Intensive Care on nurses' perspectives and decision-making skills. The study is a semi-experimental and qualitative research conducted using a single-group pre-test/post-test design.

The study consists of two phases. The first phase involves the development of the Model-Based Care Decision Support System. The second phase aims to evaluate the impact of the developed Care Decision Support System on nurses' perspectives regarding the system and their decision-making skills. A qualitative research method will be used to determine nurses' views on the Care Decision Support System, and a single-group pre-test/post-test semi-experimental design will be used to assess the effect of the decision support system on nurses' clinical decision-making skills.

The population of the study will consist of 38 nurses working in the Pediatric Intensive Care Unit of a university hospital located in the city center of Ankara. A sampling method will not be used in this study; instead, the study group will consist of nurses who meet the inclusion criteria and voluntarily agree to participate in the study.

Phase One - Development of the Care Decision Support System In this phase, a Model-Based Nursing Care Decision Support System will be developed. The system will be based on the Family-Centered Care Model and Watson's Theory of Human Caring, as these aspects of care are often overlooked in pediatric intensive care units due to the high demands of physical care. The Family-Centered Care Model emphasizes principles such as respecting the child and family (including their ethnic, cultural, socioeconomic, and racial characteristics, as well as their coping mechanisms), recognizing and supporting the strengths of the family, guiding families by supporting their preferences and decisions through care approaches, and ensuring that policies align with the family's cultural values and beliefs. Watson's Theory of Human Caring includes three main components: interpersonal caring relationships, the caring moment, and the healing processes. The nursing care components to be included in the decision support system will be identified through a qualitative study involving nurses working in pediatric intensive care units. Using the snowball sampling method, in-depth individual interviews will be conducted with nurses who are not part of the main study population. These interviews will explore which nursing care interventions should be integrated into the system. Nurses participating in this phase will be purposively selected based on criteria such as clinical experience and educational background. Pediatric intensive care nurses known to the researcher through personal or professional networks will be invited to participate. Interviews will be conducted at a suitable time outside working hours using digital platforms (e.g., Zoom, Google Meet). Data collected from these interviews will be analyzed using content analysis, and the nursing interventions to be included in the system will be finalized. Following this, the care content for the Decision Support System will be created. Expert opinion (from academic and clinical pediatric nursing professionals) will be sought to finalize the interventions to be included in the system. A software company will then be commissioned to develop the digital interface. The Care Decision Support System will incorporate the nursing process and will support nurses in identifying nursing diagnoses and selecting appropriate interventions based on patient data. The system will begin with the data collection phase of the nursing process. It will guide nurses on which data should be collected, provide alerts and prompts during analysis, and assist in clustering data to suggest possible nursing diagnoses. If a nurse selects a diagnosis but patient data is incomplete, the system will issue an alert and prompt for missing data, thereby assisting the nurse in the data analysis process. After a diagnosis is confirmed, the system will offer a set of care interventions associated with that diagnosis. Similarly, in the evaluation phase, the system will guide nurses on which outcomes should be assessed.

This comprehensive system, encompassing data collection, diagnosis, implementation, and evaluation phases of the nursing process, is designed to support pediatric intensive care nurses in making accurate care decisions. Once the software is complete, a pilot test will be conducted to assess usability and clarity. The pilot will be carried out with nurses not included in the main study sample. Necessary adjustments will be made based on the pilot, and the second phase of the study will then begin.

Phase Two - Implementation of the Care Decision Support System In this phase, data will be collected using the Descriptive Information Form, the Nurse Decision-Making Scale (as a pre-test), and the Semi-Structured Interview Form designed to explore nurses' views regarding the Decision Support System. Training will be provided to the nurses on how to use the Decision Support System, which was developed for use in providing continuous 24-hour nursing care for pediatric patients. To ensure participation, training sessions will be conducted in two groups, aligning with the nurses' work shifts so as not to disrupt clinical operations. The training will consist of two sessions totaling four hours. Topics covered will include the importance and use of the clinical decision support system, potential challenges, and suggested solutions. The system will then be introduced to the sample nurses (who meet the inclusion criteria) through hands-on application. Before full implementation in the clinical setting, a one-week trial period will be conducted to address any questions nurses may have about using the system. During this trial, the researcher will respond to all usage-related questions. A WhatsApp group including the participating nurses and the researcher will also be created to provide support throughout the implementation period.

Nurses will be required to use the system for a minimum of 15 days. Due to the time limitations of the doctoral dissertation, the maximum usage period will be 30 days. Fifteen days after the implementation ends, the post-test will be conducted using the Nurse Decision-Making Scale and a Semi-Structured Interview Form designed to evaluate the effectiveness and possible improvements of the Model-Based Nursing Care Decision Support System.

ELIGIBILITY:
Inclusion Criteria:

* Nurses with at least 6 months of experience in intensive care
* Nurses actively involved in direct patient care
* Nurses who voluntarily agree to participate in the study

Exclusion Criteria:

* Nurses who are temporarily on leave due to reasons such as maternity leave or unpaid leave

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-12-09 (Estimated); Primary Completion 2026-04-25 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Nurse Decision-Making Scale | two week
  The scale was developed by Lauri and Salanterä in 2002 . The Turkish version's validity and reliability study was conducted by Demir and Yılmaz in 2021. The scale consists of 24 items and is unidimensional. It is rated on a five-point Likert scale: "Always-5, Frequently-4, Sometimes-3, Rarely-2, Never-1." The total score ranges from 24 to 120, with higher scores indicating better decision-making skills. The Cronbach's alpha coefficient of the original scale was .84 , while it was found to be .97 in the Turkish version.

SECONDARY OUTCOMES:
Semi-Structured Interview Form for the Implementation of the Decision Support System | two week
  This form was also prepared by the researchers and finalized in line with expert feedback. It will be used twice-before and after the implementation of the Decision Support System. The form includes four open-ended questions designed to assess nurses' opinions on the system. The post-implementation version focuses specifically on evaluating the effectiveness and potential improvements of the system.

CONTACTS AND LOCATIONS:
Overall Officials: Bedriye AK, Associate Prof. Dr., Study Director — Bolu Abant İzzet Baysal Üniversity; Merve Erdem, Lecturer, Principal Investigator — Ankara Üniversity
Locations (1):
- Ankara Üniversity, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
We will prepare the study as a thesis and then publish it in an international scientific journal.
Supporting Information: Study Protocol

REFERENCES:
- [Result] Zhao Y, Hu J, Gu Y, Wan Y, Liu F, Ye C, Zhang X. Development and Implementation of a Pediatric Nursing-Clinical Decision Support System for Hyperthermia: A Pre- and Post-test. Comput Inform Nurs. 2021 Aug 4;40(2):131-137. doi: 10.1097/CIN.0000000000000812. PMID 34347639
- [Result] Tripathi, K. P. Decision support system is a tool for making better decisions in the organization. Indian Journal of Computer Science and Engineering (IJCSE),2021: 2(1), 112-117
- [Result] Demir Ş, Akman Yılmaz A. Hemşire Karar Verme Ölçeğinin Türkçeye uyarlanması: geçerlik ve güvenirlik çalışması. Sağlık ve Hemşirelik Yönetimi Dergisi. 2021;8(3):407-417.
- [Result] Lauri S, Salantera S. Developing an instrument to measure and describe clinical decision making in different nursing fields. J Prof Nurs. 2002 Mar-Apr;18(2):93-100. doi: 10.1053/jpnu.2002.32344. PMID 11977007